CLINICAL TRIAL: NCT03186742
Title: Effects of Eplerenone on Left Ventricular Hypertrophy in Patients With Resistant Hypertension and Obstructive Sleep Apnoea
Brief Title: Reduction of Left Ventricular Hypertrophy After Eplerenone Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Beata Krasinska, Principal Investigator, Poznan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 565/14
Record Dates: First submitted 2017-06-10; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Hypertension,Essential; Obstructive Sleep Apnea; Left Ventricular Hypertrophy
Keywords: Eplerenone; Concentric hypertrophy
MeSH Terms: conditions — Essential Hypertension; Sleep Apnea, Obstructive; Hypertrophy, Left Ventricular | interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): The patients who had Eplerenone 50mg tab once a day added to their standard hypertensive treatment.
  Interventions: Drug: Eplerenone 50 mg Tab
- Group B (No Intervention): The patients who did not receive an additional drug to their standard hypertensive treatment.

INTERVENTIONS:
Drug: Eplerenone 50 mg Tab — Eplerenone 50 mg Tab once a day
  Arms: Group A

SUMMARY:
Obstructive sleep apnea syndrome (OSA) is the most frequent sleep disorder characterized by excessive decrease in muscle tone of the soft palate, the tongue and the posterior pharyngeal wall. It leads to airway collapse. In cases of decreased airway passage hypoventilation (hypopnea) occurs while periodic lack of airflow is called apnea. An obstructive sleep apnea syndrome is recognized as an independent cardiovascular risk factor. OSA is very common in patients with resistant hypertension. RAH is diagnosed when blood pressure remains elevated despite simultaneous use of 3 antihypertensive agents from different groups of drugs at optimal to maximum doses, including a diuretic.

In patients with OSA frequent episodes of hypoxemia during sleep result in the repeated activation of the sympathetic nervous system. What is more, the episodes of respiratory disorders increases in levels of aldosterone serum concentration with following sodium and water retention and elevation of blood pressure finally. An increased aldosterone level also stimulates synthesis of collagen, promotes stiffening of the arterial wall, myocardial fibrosis with heart muscle remodeling and takes part in development of left ventricular hypertrophy (LVH) - common complication of hypertensive patients with OSA. Several studies, including the Sleep Heart Health Study have confirmed that severe OSA is associated with high prevalence of concentric hypertrophy through sympathetic activation and vasoconstriction.

Eplerenone is a selective mineralocorticoid receptor inhibitor. It has no affinity for glucocorticoid, progesterone and androgen receptors and therefore has lower risk of side effects. Eplerenone lowers blood pressure and inhibits heart muscle fibrosis. The hypotensive effect is caused by reduction of fluid retention. Probably, in patients with OSA, a reduction of fluid accumulation especially at the level of the neck may contribute to lowering the resistance in the upper respiratory tract and in that way it may help to decrease the severity of OSA.

As LVH remains a strong and independent predictor of total mortality and death from cardiovascular causes, in this study we want to assess whether the addition of Eplerenone to a standard antihypertensive therapy will favorably change left ventricular geometry. We also want to check if the addition the Eplerenone to a standard antihypertensive therapy could be an effective therapeutic option for patients with OSA and RAH.

DETAILED DESCRIPTION:
125 patients (78 men and 47 women) aged 18 - 65 years, with diagnosed resistant hypertension and moderate or severe OSA were included in the study, which was conducted in years 2014-2017 in the Department of Hypertension, Angiology and Internal Medicine and the Department of Pulmonology, Allergology and Respiratory Oncology at the University of Medical Sciences in Poznan, Poland. 23 patients did not complete the study because they did not meet the inclusion criteria (10 patients) and did not follow the recommendations (13 patients). 102 patients were randomized to two groups. In Group A, 50mg Eplerenone was administered orally once a day additionally for standard antihypertensive therapy. In Group B, standard antihypertensive therapy was not changed for 6 months of follow-up. RAH was recognized when in spite of the use of at least 3 antihypertensive agents (including a diuretic) in maximum doses, it was impossible to achieve the target values of BP (< 140/90 mmHg). The patients were taking on average 3,93 antihypertensive medications including diuretics (100% of patients), angiotensin-converting enzyme inhibitors (54% of patients), angiotensin II receptor antagonists (45.2% of patients), calcium antagonists (83.9% of patients), β-blockers (77.4% of patients), and α-blockers (22.6% of patients). The permission no. 565/14 to conduct the study was granted by the Ethics Committee of the University of Medical Sciences in Poznan. All patients gave an informed and written consent to participation in the study. Blood pressure measurements In all patients, during each visit, BP measurements were performed three times at rest in supine position, in standard conditions, using an upper arm blood pressure monitor BP monitor (Omron 705IT, Omron Healthcare, Kyoto, Japan). Ambulatory 24-hours BP automated monitoring (ABPM) was performed using a 24-hour ambulatory peripheral BP monitor TM2430 (A&D Medical, San Jose, California, United States). The frequency of measurements was every 15 minutes between 7:00 and 22:00 and every 30 minutes between 22:00 and 7:00.

Neck circumference measurement The neck circumference was measured in the midway of the neck, between the mid-cervical spine and mid-anterior neck, in standing position, with a flexible no-stretchable plastic tape, and approximated to the nearest 0.1 cm.

Echocardiographic examination

All patients underwent complete transthoracic echocardiographic study with Vivid S6 (GE Medical System, Tirat Carmel, Israel) with a 1,5 - 3,6 megahertz cardiac sector probe. A standard M-mode, two-dimensional and Doppler echocardiographic examination was performed according to the guidelines of American Society of Echocardiography. Three consecutive cycles were averaged for every parameter. The same experienced cardiologist who was blinded to the presence or absence of OSA performed all echocardiographic examinations. Left ventricular end-diastolic diameter (LVED), thickness of intraventricular septum at end diastole (IVS), left ventricular posterior wall at end diastole (LVPW) and left ventricular mass (LVM) were measured according to American Society of Echocardiography recommendations. The LVH was defined as the IVS or the LVPW>12 mm. The left ventricular mass was calculated using a simple and anatomically validated formula:

LVM = 0.8 × 1.04 [(IVS + LVED + LVPW) 3 - LVED 3] + 0.6 LVM was calculated as corrected for height and LVM index (LVMI). The relative wall thickness (RWT) was calculated as (2× LVPW)/LVEDD, for which the normal limit is <0.42. Based on LVMI and RWT, the LV geometry was classified as normal (LVMI <115 g/m2 in men, <95 g/m2 in women and RWT <0.42), concentric remodeling (normal LVMI <115 g/m2 in men, <95 g/m2 in women and increased RWT >0.42), concentric hypertrophy (LVMI >115 g/m2 in men, >95 g/m2 in women and increased RWT >0.42) or eccentric hypertrophy (LVMI >115 g/m2 in men, >95g/m2 in women and normal RWT <0.42).

Polysomnography (PSG) The probability of OSA was established at first on the base of Epworth Sleepiness Scale score. The evaluation of patients was performed in the Sleep Laboratory of the Department of Pulmonology, Allergology and Respiratory Oncology at the University of Medical Sciences in Poznan, Poland using a full-night polysomnographic monitoring system (EMBLA S4000, Remlogic, Denver, Colorado) with Somnologica studio 3.3.2 software (EMBLA, Broomfield, Colorado, United States). Standard electroencephalography monitoring, including frontal leads (F1, F2), central leads (C3, C4), occipital leads (O1, O2) and reference leads at the mastoids (M1, M2); electromyography and electrooculography methodology were performed according to The American Academy of Sleep Medicine (AASM) guidelines.

Airflow was measured using nasal thermistors, and a nasal pressure transducer. Abdominal and thoracic movements were assessed by respiratory inductive plethysmography. Oximetry was measured using a disposable finger probe (oximeter flex sensor 8000 J, NONIN, Plymouth, Massachusetts, United States) placed on the index finger. Snoring sounds, heart rate also were recorded. Body position was monitored using body position sensor. Apnea was defined as a cessation of airflow lasting for more than 10 sec., and hypopnea as a discrete reduction (two thirds) of airflow and/or abdominal ribcage movements lasting for more than 10 sec. and associated with a decrease of more than 4% in oxygen saturation. Trained PSG technicians and sleep physicians using the criteria of Rechtschaffen and Kales, and in close concordance with scoring updates given by the American Academy of Sleep Medicine analyzed all studies. The apnea-hypopnea index (AHI) was defined by the total number of apneas and hypopneas per hour of sleep. The severity of OSA was determined as: mild (AHI 5-15), moderate (AHI 15 - 30) and severe (AHI ≥ 30) (21) on the basis of AHI Design of the study First visit Patients with previously diagnosed RAH and with suspected OSA (medical history, the Epworth scale assessment) were referred from an outpatient clinic to the hospital ward. After admission numerous laboratory tests and imaging, such as aldosterone and Plasma renin activity levels (ARO), both before and after tilting, creatinine, urea, GFR, sodium and potassium levels, pro B-type natriuretic peptide (BNP), thyrotrophin (TSH), free triiodothyronine (FT3), free thyroxine(fT4), 24-hour urine collection for electrolytes, as well as abdominal ultrasound examinations, computed tomography of the abdomen and Doppler ultrasound of the renal arteries, were performed to exclude secondary causes of arterial hypertension (other than primary hyperaldosteronism). What is more, office BP was measured three times at admission and afterwards 24-hours ABPM examination was conducted. All participants underwent also transthoracic echocardiography. After aforementioned diagnostics and after confirming RAH based on 24-hour ABPM, patients were referred to the Department of Pulmonology to perform polysomnography.

In those patients in who moderate or severe OSA (AHI>15/h), had been confirmed, Eplerenone at the dose of 50 mg/day was randomly added to the previously used treatment regimen.

Second visit After six months, office BP (measured three times in standard conditions as initially performed), 24-hour ABPM, echocardiography and polysomnography were repeated.

Statistical analysis The normality of distribution of the analyzed variables was evaluated with the Shapiro-Wilk test and Kolmogorov-Smirnov test with the Lilliefors correction. The results of the tests showed that distributions of almost all parameters significantly differed from the normal distribution. Therefore, nonparametric methods were used in statistical analysis. The Wilcoxon signed-rank test was applied for the evaluation of the differences between the baseline values and those obtained after treatment. The t test was used for variables with normal distribution. Correlations between the values of the parameters were evaluated using the Spearman's rank correlation coefficient. P value of less than 0.05 was considered significant. The Statistica software, version 10, was used for the analysis (www. statsoft. com; license JGNP410B316631AR-J, Stat- Soft, Inc., 2011, Tulsa, Oklahoma, United States).

ELIGIBILITY:
Inclusion Criteria:

* confirmation of resistant hypertension(RAH). RAH was recognized when in spite of the use of at least 3 antihypertensive agents (including a diuretic) in maximum doses, it was impossible to achieve the target values of BP (< 140/90 mmHg).
* diagnosing of moderate or severe sleep apnea (OSA) on the basis of apnoea-hypopnea index (AHI) in polysomnography. AHI was defined by the total number of apnoea's and hypopneas per hour of sleep. The severity of OSA was determined as: mild (AHI 5-15), moderate (AHI 15 - 30) and severe (AHI ≥ 30)
* signing informed and written consent to participation in the study.

Exclusion Criteria:

* secondary hypertension (other than primary hyperaldosteronism),
* myocardial infarction,
* stroke within 6 months before the study,
* congestive heart failure with New York Heart Association (NYHA) grade III-IV,
* chronic kidney disease (GFR < 30 ml/min),
* active addiction to alcohol or psychoactive substances,
* active cancer disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with reduction of left ventricular hypertrophy after Eplerenone therapy | 6 months
  Changes in echocardiographic data ( LVED, IVS, LVPW, LVMI, RWT) and in left ventricular geometric patterns after six months Eplerenone treatment

SECONDARY OUTCOMES:
Reduction in blood pressure after Eplerenone therapy | 6 months
  Reduction in office BP (measured three times in standard conditions) and in 24-hour ABPM parameters
Reduction in (AHI) apnea-hypopnea index after Eplerenone therapy | 6 months
  AHI - parameter determining the severity of OSA in polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Tykarski, Prof, Study Chair — Department of Hypertension, Angiology and Internal Disease. Poznan University of Medical Sciences, Poland; Szczepan Cofta, PhD, Principal Investigator — Department of Respiratory Diseases, Allergology and Lung Oncology. Poznan University of Medical Sciences, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sleep-related breathing disorders in adults: recommendations for syndrome definition and measurement techniques in clinical research. The Report of an American Academy of Sleep Medicine Task Force. Sleep. 1999 Aug 1;22(5):667-89. No abstract available. PMID 10450601
- [Result] Lavie P, Herer P, Hoffstein V. Obstructive sleep apnoea syndrome as a risk factor for hypertension: population study. BMJ. 2000 Feb 19;320(7233):479-82. doi: 10.1136/bmj.320.7233.479. PMID 10678860
- [Result] Shahar E, Whitney CW, Redline S, Lee ET, Newman AB, Nieto FJ, O'Connor GT, Boland LL, Schwartz JE, Samet JM. Sleep-disordered breathing and cardiovascular disease: cross-sectional results of the Sleep Heart Health Study. Am J Respir Crit Care Med. 2001 Jan;163(1):19-25. doi: 10.1164/ajrccm.163.1.2001008. PMID 11208620
- [Result] ESH/ESC Task Force for the Management of Arterial Hypertension. 2013 Practice guidelines for the management of arterial hypertension of the European Society of Hypertension (ESH) and the European Society of Cardiology (ESC): ESH/ESC Task Force for the Management of Arterial Hypertension. J Hypertens. 2013 Oct;31(10):1925-38. doi: 10.1097/HJH.0b013e328364ca4c. No abstract available. PMID 24107724
- [Result] Drager LF, Bortolotto LA, Figueiredo AC, Silva BC, Krieger EM, Lorenzi-Filho G. Obstructive sleep apnea, hypertension, and their interaction on arterial stiffness and heart remodeling. Chest. 2007 May;131(5):1379-86. doi: 10.1378/chest.06-2703. PMID 17494787
- [Result] Cioffi G, Russo TE, Stefenelli C, Selmi A, Furlanello F, Cramariuc D, Gerdts E, de Simone G. Severe obstructive sleep apnea elicits concentric left ventricular geometry. J Hypertens. 2010 May;28(5):1074-82. doi: 10.1097/hjh.0b013e328336c90a. PMID 20411620
- [Result] Chami HA, Devereux RB, Gottdiener JS, Mehra R, Roman MJ, Benjamin EJ, Gottlieb DJ. Left ventricular morphology and systolic function in sleep-disordered breathing: the Sleep Heart Health Study. Circulation. 2008 May 20;117(20):2599-607. doi: 10.1161/CIRCULATIONAHA.107.717892. Epub 2008 May 5. PMID 18458174
- [Result] Alchanatis M, Paradellis G, Pini H, Tourkohoriti G, Jordanoglou J. Left ventricular function in patients with obstructive sleep apnoea syndrome before and after treatment with nasal continuous positive airway pressure. Respiration. 2000;67(4):367-71. doi: 10.1159/000029532. PMID 10940788
- [Result] Yamaguchi T, Takata Y, Usui Y, Asanuma R, Nishihata Y, Kato K, Shiina K, Yamashina A. Nocturnal Intermittent Hypoxia Is Associated With Left Ventricular Hypertrophy in Middle-Aged Men With Hypertension and Obstructive Sleep Apnea. Am J Hypertens. 2016 Mar;29(3):372-8. doi: 10.1093/ajh/hpv115. Epub 2015 Jul 23. PMID 26208670
- [Result] Gaddam K, Pimenta E, Thomas SJ, Cofield SS, Oparil S, Harding SM, Calhoun DA. Spironolactone reduces severity of obstructive sleep apnoea in patients with resistant hypertension: a preliminary report. J Hum Hypertens. 2010 Aug;24(8):532-7. doi: 10.1038/jhh.2009.96. Epub 2009 Dec 17. PMID 20016520
- [Result] Struthers A, Krum H, Williams GH. A comparison of the aldosterone-blocking agents eplerenone and spironolactone. Clin Cardiol. 2008 Apr;31(4):153-8. doi: 10.1002/clc.20324. PMID 18404673
- [Result] Lorell BH, Carabello BA. Left ventricular hypertrophy: pathogenesis, detection, and prognosis. Circulation. 2000 Jul 25;102(4):470-9. doi: 10.1161/01.cir.102.4.470. No abstract available. PMID 10908222
- [Result] Schiller NB, Shah PM, Crawford M, DeMaria A, Devereux R, Feigenbaum H, Gutgesell H, Reichek N, Sahn D, Schnittger I, et al. Recommendations for quantitation of the left ventricle by two-dimensional echocardiography. American Society of Echocardiography Committee on Standards, Subcommittee on Quantitation of Two-Dimensional Echocardiograms. J Am Soc Echocardiogr. 1989 Sep-Oct;2(5):358-67. doi: 10.1016/s0894-7317(89)80014-8. PMID 2698218
- [Result] Devereux RB, Alonso DR, Lutas EM, Gottlieb GJ, Campo E, Sachs I, Reichek N. Echocardiographic assessment of left ventricular hypertrophy: comparison to necropsy findings. Am J Cardiol. 1986 Feb 15;57(6):450-8. doi: 10.1016/0002-9149(86)90771-x. PMID 2936235
- [Result] Lang RM, Bierig M, Devereux RB, Flachskampf FA, Foster E, Pellikka PA, Picard MH, Roman MJ, Seward J, Shanewise JS, Solomon SD, Spencer KT, Sutton MS, Stewart WJ; Chamber Quantification Writing Group; American Society of Echocardiography's Guidelines and Standards Committee; European Association of Echocardiography. Recommendations for chamber quantification: a report from the American Society of Echocardiography's Guidelines and Standards Committee and the Chamber Quantification Writing Group, developed in conjunction with the European Association of Echocardiography, a branch of the European Society of Cardiology. J Am Soc Echocardiogr. 2005 Dec;18(12):1440-63. doi: 10.1016/j.echo.2005.10.005. No abstract available. PMID 16376782
- [Result] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Result] Smith SS, Oei TP, Douglas JA, Brown I, Jorgensen G, Andrews J. Confirmatory factor analysis of the Epworth Sleepiness Scale (ESS) in patients with obstructive sleep apnoea. Sleep Med. 2008 Oct;9(7):739-44. doi: 10.1016/j.sleep.2007.08.004. Epub 2007 Oct 24. PMID 17921053
- [Result] Hori T, Sugita Y, Koga E, Shirakawa S, Inoue K, Uchida S, Kuwahara H, Kousaka M, Kobayashi T, Tsuji Y, Terashima M, Fukuda K, Fukuda N; Sleep Computing Committee of the Japanese Society of Sleep Research Society. Proposed supplements and amendments to 'A Manual of Standardized Terminology, Techniques and Scoring System for Sleep Stages of Human Subjects', the Rechtschaffen & Kales (1968) standard. Psychiatry Clin Neurosci. 2001 Jun;55(3):305-10. doi: 10.1046/j.1440-1819.2001.00810.x. No abstract available. PMID 11422885